CLINICAL TRIAL: NCT01360736
Title: A Brief Intervention to Reduce Suicide Risk in Military Service Members and Veterans - Study 2
Brief Title: A Brief Intervention to Reduce Suicide Risk in Military Service Members and Veterans - Study 2 (SAFEMIL)
Acronym: SAFEMIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency); University of Pennsylvania (Other); University of Rochester (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Marjan Holloway, Principal Investigator (Contact PI), Henry M. Jackson Foundation for the Advancement of Military Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-09-2-0129 Study 2
Record Dates: First submitted 2011-05-17; First posted 2011-05-26 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Suicide; Suicide, Attempted
Keywords: Suicide Prevention; Suicide Attempt; Suicide Ideation; Randomized Controlled Trial; Safety Planning
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicide Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Safety Planning - Military (SAFE-MIL) (Experimental): Brief Safety Planning Using Stanley and Brown (2012) Model
  Interventions: Behavioral: Safety Planning - Military (SAFE MIL)
- E-CARE (No Intervention): Treatment As Usual and Assessment Services of Study; Control Condition

INTERVENTIONS:
Behavioral: Safety Planning - Military (SAFE MIL) — The Safety Planning Intervention (SPI) which is delivered in the SAFE MIL condition aims to help individuals lower their imminent suicide risk by having them collaborate with the study clinician to generate a detailed, hierarchically-arranged action plan for managing suicidal thoughts and urges.
  Other Names: Safety Planning
  Arms: Safety Planning - Military (SAFE-MIL)

SUMMARY:
The investigators propose to test the efficacy of a brief, readily accessible, and personalized treatment called the Safety Planning for Military (SAFE MIL; Stanley and Brown, 2012).

DETAILED DESCRIPTION:
Background: Mental health related hospitalizations and suicide are both significant public health problems within the United States Department of Defense (DoD). There are limited evidence-based suicide prevention interventions that have been developed for military personnel and veterans who are experiencing suicide ideation or who have made a suicide attempt.

Objectives: To evaluate the efficacy of the Safety Planning for Military (SAFE MIL) on suicide ideation, suicide-related coping, and attitudes toward help seeking for hospitalized military personnel at high suicide risk.

Methodology: To test the efficacy of the adapted intervention, the investigators will randomize 186 patients to one of two conditions: Safety Planning for Military (SAFE MIL) or Enhanced Usual Care (E-CARE). The SAFE MIL condition (intervention) will consist of the Safety Planning Intervention to help the suicidal individual with a collaboratively generated personal plan to mitigate or prevent a future suicidal crisis. The E-Care will consist of the usual care patients receive at an inpatient facility during their hospitalization in addition to assessment services provided by independent evaluators who work directly with our research team. Primary outcomes include suicide ideation, suicide-related coping, and attitudes toward help-seeking [acceptability and initiation of services]. Patients in both conditions will be assessed on the dependent measures at the time of hospital admission (i.e., baseline), at the time discharge (Follow-Up Interval 1 [FU-1]), at 1-month (Follow-Up Interval 2 [FU-2]) and at 6-month (Follow-Up Interval 3 [FU-3]).

ELIGIBILITY:
Inclusion Criteria:

* Patient Admitted Due to Recent Suicide Intent and/or Suicide Attempt within past month
* Baseline Assessment Completed within 48 Hours of Hospital Admission
* Age of 18 years or older.

Exclusion Criteria:

* Medical Incapacity to Participate and/or Serious Cognitive Impairment
* Expected Discharge within 72 Hours of Admission
* Expected Deployment within 1-Month
* Inability to read or understand English
* Inability to provide Informed Consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-09; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Suicide Ideation | discharge, 1 month, and 6 months post-discharge
  Suicide ideation will be measured using the Columbia Suicide Severity Rating Scale (C-SSRS) and the Scale for Suicide Ideation (SSI). Both measures assess for presence, intensity, frequency, and specificity of suicide related thoughts (ideations).
Acceptability and Initiation of Mental Health Care and Substance Use Treatment | discharge, 1 month, and 6-months post-discharge
  Attitudes toward help-seeking [acceptability and initiation of services] will be assessed by the following measures: Attitudes Toward Seeking Professional Psychological Help Scale: modified shortened version (ATSPPH); Cornell Services Index (CSI); Perceived Barriers to Care (PBTC); Brief SAFE MIL Intervention Survey.
Suicide-related Coping | discharge, 1 month, and 6 months post-discharge
  Coping strategies will be measured using a checklist of tactics and coping strategies used by individuals to cope with suicidal thoughts, feelings, and urges.

CONTACTS AND LOCATIONS:
Overall Officials: Marjan G Holloway, Ph.D., Principal Investigator — Uniformed Services University of the Health Sciences; Lisa Brenner, Ph.D., Principal Investigator — Denver VA; Gregory Brown, Ph.D., Principal Investigator — University of Pennsylvania; Glenn Currier, M.D., MPH, Principal Investigator — Canandaigua VA; University of Rochester; Kerry Knox, Ph.D., Principal Investigator — Canandaigua VA; University of Rochester; Barbara Stanley, Ph.D., Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Uniformed Services University of the Health Sciences, Bethesda, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knox KL, Stanley B, Currier GW, Brenner L, Ghahramanlou-Holloway M, Brown G. An emergency department-based brief intervention for veterans at risk for suicide (SAFE VET). Am J Public Health. 2012 Mar;102 Suppl 1(Suppl 1):S33-7. doi: 10.2105/AJPH.2011.300501. PMID 22390597
- [Background] Ghahramanlou-Holloway M, Brown GK, Currier GW, Brenner L, Knox KL, Grammer G, Carreno-Ponce JT, Stanley B. Safety Planning for Military (SAFE MIL): rationale, design, and safety considerations of a randomized controlled trial to reduce suicide risk among psychiatric inpatients. Contemp Clin Trials. 2014 Sep;39(1):113-23. doi: 10.1016/j.cct.2014.07.003. Epub 2014 Jul 12. PMID 25020008